CLINICAL TRIAL: NCT02248025
Title: Can Capillary Refill Time Variation Induced by Passive Leg Raising Predict Capillary Refill Time Variation After a Fluid Load in Patients With Circulatory Failure.
Brief Title: Can Capillary Refill Time Variation During Passive Leg Raising Predict Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Hopital Louis Pradel (Other)
Responsible Party: Principal Investigator, Matthias Jacquet-Lagrèze, Dr Matthias Jacquet-Lagèze, Hopital Louis Pradel
Other Study IDs: EudraCT/ANSM: 2014-A01034-43
Record Dates: First submitted 2014-09-13; First posted 2014-09-25 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Circulatory Failure
Keywords: Fluid responsiveness; capillary refill time; microcirculation; circulatory failure; passive leg raising
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study: No special intervention will be made. — No special intervention will be made, only data will be collected before, and after a passive leg raising and a fluid challenge decided and performed by the attending physician.

SUMMARY:
Fluid responsiveness in a context of circulatory failure can be assessed by different way. Microcirculatory evaluation to assess fluid responsiveness could be interesting, but the available device are expensive and the analysis are delayed. Capillary refill time (CRT) is hampered by its variability. The investigators have developed a method to standardize the pressure, the length of compression and a computerized analysis to calculate the capillary refill time. This method enables accurate measure of CRT.

The investigators will study if CRT variation induced by a passive leg raising (PLR) can predict CRT after a 500 ml Fluid Load.

About thirty patients in circulatory failure with a continuous cardiac output monitoring for whom, the attending physician has decided a fluid load, will be included. hemodynamic parameters (arterial pressure, venous pressure, cardiac output), metabolic parameters (arterial and venous blood gas and lactate), microcirculatory parameters (assessed by sublingual video-microscopy) and capillary refill time measured on the thorax and on the gingival area will be recorded. Data collection will be made before and after a passive leg raising and after a 500 ml fluid load of crystalloids.

Patients will be aposteriori sorted in two groups: responders and non responders, defined by the reduction of CRT after the fluid load. The diagnosis ability of the CRT variation after PLR to predict in which group each patient is classified will be investigate and receiver operative characteristic curve will be built. These results will be compared to the metabolic response, the macrocirculatory response, and the microcirculatory response.

ELIGIBILITY:
Inclusion Criteria:

* The patient is equipped with an arterial and a central venous catheter
* Capillary refill time is measurable.
* A cardiac output monitoring is available
* A 500 ml fluid load as been prescribed by the intensivist in charge.
* A circulatory failure is present defined as follow:

Patient treated with inotropic or vasoconstrictive drugs

OR

Patient presenting an hypotension defined by systolic arterial pressure less than 90 mmHg or mean arterial pressure less than 70 mmHg or a drop 40 mmHg in case of previous Hypertension.

WITH

tissue hypoperfusion defined by at least one of the following item:

* Lactate > 1 mmol/L
* Capillary refill time > 3 s
* Blotch
* Organ dysfunction due to the circulatory failure (oligo anuria, acute lung injury / acute respiratory distress syndrome, encephalopathy)

Exclusion Criteria:

* Pregnant woman
* Cardiogenic pulmonary edema
* Circulatory support : extracorporal life support / extracorporal membrane oxygenator, Thoratec, heart mate.
* Moribund patient
* Intra-abdominal hypertension
* Lower limb amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in our intensive care unit who are in circulatory failure and for whom the intensivist as decided to administer a 500 ml crystalloid infusion.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Capillary refill time response | The period of inclusion last 45 minutes, the outcome will be assessed at the end of the 500 ml fluid load 45 minutes after the inclusion.
  A reduction of about 30% of the capillary refill time after a 500 ml fluid load will defined responders.
  Evaluation of the diagnosis capacity of capillary refill time variation after passive leg raising to diagnose responders will be investigate.

SECONDARY OUTCOMES:
Cardiac output response. | The period of inclusion last 45 minutes, the outcome will be assessed at the end of the 500 ml fluid load 45 minutes after the inclusion.
  An increase of 15% of cardiac output after a 500 ml fluid load will define macrocirculatory responders.
  Evaluation of the diagnosis capacity of capillary refill time after passive leg raising to diagnose macrocirculatory responders will be investigate.
Microcirculatory response | The period of inclusion last 45 minutes, the outcome will be assessed at the end of the 500 ml fluid load 45 minutes after the inclusion.
  An increase of 15% of the proportion of perfused vessels or from 0.6 of the microcirculatory flow index assessed by videomicroscopy after a 500 ml fluid load will define microcirculatory responders.
  Evaluation of the diagnosis capacity of capillary refill time variation after passive leg raising to diagnose microcirculatory responders will be investigate.
Metabolic response | The period of inclusion last 45 minutes, the outcome will be assessed at the end of the 500 ml fluid load 45 minutes after the inclusion.
  An increase of 15% Oxygen consumption after a 500 ml fluid load will define metabolic responders.
  Evaluation of the diagnosis capacity of capillary refill time to diagnose metabolic responders after passive leg raising will be investigate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cardiologique Louis Pradel Service d'anesthésie réanimation, Bron, France

REFERENCES:
- [Derived] Jacquet-Lagreze M, Bouhamri N, Portran P, Schweizer R, Baudin F, Lilot M, Fornier W, Fellahi JL. Capillary refill time variation induced by passive leg raising predicts capillary refill time response to volume expansion. Crit Care. 2019 Aug 16;23(1):281. doi: 10.1186/s13054-019-2560-0. PMID 31420052